CLINICAL TRIAL: NCT00973102
Title: Resuscitative Endocrinology: (RESCUE - Shock): A Phase II Trial to Evaluate the Effects of Single Dose Intravenous Premarin for Treatment of Patients With Hemorrhagic Shock
Brief Title: Resuscitative Endocrinology: Single-dose Clinical Uses for Estrogen-Traumatic Hemorrhagic Shock (RESCUE - Shock)
Acronym: RESCUE-Shock
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: University of Washington (Other); Resuscitation Outcomes Consortium (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RESCUE - Shock
Record Dates: First submitted 2009-07-19; First posted 2009-09-09 (Estimated); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Hemorrhagic Shock
MeSH Terms: conditions — Shock, Hemorrhagic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Premarin IV (Experimental): Patients who were randomized to receive a single dose of 0.5 mg/kg Premarin® IV.
  Interventions: Drug: Premarin IV
- Placebo (Placebo Comparator): Patients who were randomized to receive a single dose of 0.5 mg/kg placebo. Due of the faint yellow color of the reconstituted Premarin®, the placebo dose will be prepared with 0.14 ml of Vial 1 of Infuvite Adult Multivitamin and 14 ml of sterile water to generate a similar color and volume. This aliquot will be used only for those study patients who are randomized to the placebo arm. The placebo volume will be approximately equal to the volume which the patient would have received had the patient been randomized to the Premarin arm Considering the small amount of IV multivitamin needed for fluid tinting, it is not expected that the IV multivitamin will have any effect on patients with hemorrhagic shock.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Premarin IV — One time dose of Premarin IV
  Other Names: Estrogen IV
  Arms: Premarin IV
Drug: Placebo — One time dose of placebo.
  Other Names: Infuvite Multivitamin
  Arms: Placebo

SUMMARY:
Based on encouraging results from animal studies, the investigators hypothesize that early administration of IV Premarin® in patients with hemorrhagic shock will safely reduce secondary injury, and improve survival.

DETAILED DESCRIPTION:
Annually in the United States, approximately 30 million people require treatment for traumatic injuries in emergency departments. Two million of these patients require hospitalization, with several hundred thousand ultimately dying, often due to extreme blood loss. Importantly, these traumatic injuries are the leading cause of death and disability for children and young adults under the age of 44, with the total cost of trauma in the U.S. approaching $260 billion each year.

Despite advances in pre-hospital care, early resuscitation, surgical interventions and intensive care monitoring aimed at the primary traumatic injury, many survivors never recover. A significant cause of this mortality and morbidity is thought due to potentially preventable secondary injury, namely oxidant injury, inflammation, and apoptosis beginning in the first few hours after the severe traumatic event.

In spite of the current bleak outlook for many of these patients, a series of animal investigations have uncovered a promising solution to the problem of the secondary injury seen in hemorrhagic shock and other similar processes, namely the early administration of estrogen, a strong anti-oxidant, anti-inflammatory and anti-apoptotic compound.

Based on encouraging results from animal studies, the investigators hypothesize that early administration of IV Premarin® in patients with hemorrhagic shock will safely reduce secondary injury, and improve survival.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥ 18 yrs or < 50 yrs
2. Blunt or penetrating trauma leading to presumed hemorrhagic shock
3. Pre-hospital or ED systolic blood pressure < 90
4. Receiving medical treatment in the Emergency Department (ED) of Parkland Hospital or Baylor University Medical Center Emergency Department, Level I Trauma Centers in Dallas, Texas

Exclusion Criteria:

1. Those who would receive the study drug > 120 minutes after the traumatic event
2. Time of injury is unknown
3. Known indication for IV estrogen
4. Known contraindication for estrogen
5. Estimated age <18 or > 50 years
6. Cardiopulmonary Resuscitation (CPR) prior to randomization
7. Known incarceration
8. Severe hypothermia (suspected T < 28° C)
9. Drowning or asphyxia due to hanging
10. Burns total body surface area (TBSA) > 20%
11. Isolated penetrating injury to the head
12. Known inclusion in another interventional trial related to this traumatic event prior to randomization
13. Known legal do not resuscitate (DNR) orders in place prior to randomization
14. Recognized spinal cord injury prior to study drug administration

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2009-07; Primary Completion 2012-01 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rob Schmickers, Study Director — University of Washington
Locations (2):
- United States (2):
  - Parkland Hospital, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinical sites enrolled men and women age 18 to 55 who experienced hemorrhagic shock in the emergency medical services (EMS) setting between September 2009 and January 2012.
Period: Overall Study
Arm/Group | Premarin IV | Placebo
Started | 24 | 26
Completed | 23 | 25
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Prisoner | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Premarin IV | Placebo | Total
Number analyzed (Participants) | 23 | 25 | 48
Age, Continuous [Mean (Full Range); unit: years] | 33.9 [17 to 54] | 32.2 [20 to 56] | 33.0 [17 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 20 | 21 | 41
Region of Enrollment [Number; unit: participants]
  United States | 23 | 25 | 48

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: Survival is defined as the number of patients who were discharged from the hospital alive prior to 28 days post injury or the number of patients still alive in the hospital 28 days post injury. The trial examines the rate of enrolled patients on each arm who survived to 28 days.
Time Frame: 28 Days
Measure: Number; unit: participants
Arm/Group | Premarin IV | Placebo
Number analyzed (Participants) | 23 | 25
participants | 16 | 21
Statistical Analysis 1: Comparison: Premarin IV vs Placebo; Test type: Superiority or Other; p = .252, Barnard's unconditional Exact Test; Hazard Ratio (HR) = 2.47, 95% CI 2-sided [1.16 to 5.25]

2. Secondary Outcome: Acute Respiratory Distress Syndrome (ARDS) Free Survival
Description: ARDS is a life-threatening condition characterized by inflammation of the lungs. The trial measures the number of days alive and without ARDS within 28 days post injury. Patients who die within 28 days are given value of 0, similarly, patients who live 28 days but have ARDS for all 28 days. A higher score (greater days) indicates better prognosis. Exudative stage is 0-6 days, proliferative stage is 7-10 days, Fibrotic stage is >10-14 days.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Premarin IV | Placebo
Number analyzed (Participants) | 23 | 25
units on a scale | 3.00 (3.46) | 3.33 (3.01)
Statistical Analysis 1: Comparison: Premarin IV vs Placebo; Test type: Superiority or Other; p = .895, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Premarin IV | Placebo
Serious Adverse Events (participants affected / at risk) | 5/23 | 7/25
Other Adverse Events (participants affected / at risk) | 0/23 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Premarin IV (N=23) | Placebo (N=25)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bloodstream (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Line infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 2 (2) | 4 (4)
Intra-abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary embolus (Vascular disorders) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes